CLINICAL TRIAL: NCT05880576
Title: The Arch Watch Study: An Integrated Evaluation of Hemodynamics During Monitoring of Ductus Arteriosus Closure in Infants With Suspected Coarctation of the Aorta
Brief Title: The Arch Watch Study: An Integrated Evaluation of Hemodynamics in Infants With Suspected Coarctation of the Aorta
Status: Enrolling by invitation | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, John Kheir, Associate Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: P00044159
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Coarctation of the Aorta; Aortic Arch Obstruction
MeSH Terms: conditions — Aortic Coarctation | interventions — Oximetry; Blood Pressure; Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Monitoring using resonance Raman spectroscopy, pulse oximetry, blood pressure, and near-infrared spectroscopy — Infants will have monitoring three times a day with resonance Raman spectroscopy device during arch watch period. They will have continuous monitoring with pulse oximetry and near infrared spectroscopy. They will have intermittent blood pressure monitoring.

SUMMARY:
Unrecognized coarctation of the aorta (CoA) is a life-threatening component of congenital heart disease (CHD) in which narrowing of the aorta causes obstructed blood flow to the lower half of the body; it can occur in isolation or in combination with other defects. CoA is the type of CHD most likely to be missed by current newborn screening. An evolving coarctation (during closure of the ductus arteriosus) can be challenging to diagnose until often devastating end-organ injury manifests, even in the ICU setting. This study will evaluate currently used tools, such as four extremity blood pressures and pulse oximetry, and the investigators will test new tools - resonance Raman spectroscopy (RRS) and photoplethysmography analysis- to assess the adequacy of oxygen delivery in newborns who are at risk for aortic arch obstruction. The investigators hypothesize that combining an assessment of commonly used non-invasive monitoring tools, new components of these traditional tools, and RRS, will have improved sensitivity in detecting critical impairments to tissue oxygen delivery in newborns with suspected critical aortic arch obstruction.

DETAILED DESCRIPTION:
Coarctation of the aorta (CoA) is a potentially life-threatening form of congenital heart disease (CHD) in which an anatomic narrowing of the aortic arch may cause critical aortic arch obstruction (AAO) following closure of the ductus arteriosus (DA). CoA accounts for 6-8% of all CHD and occurs in about 1 in every 1800 babies born in the United States each year. Despite this prevalence, CoA frequently eludes detection on both prenatal imaging and CHD screening. If undiagnosed, infants may present with catastrophic shock, often leading to mortality or severe morbidities. In many cases, the anatomic appearance of the aortic arch in the fetal or early postnatal period raises suspicion for AAO that can only be confirmed by allowing the DA to become restrictive and closely monitoring for hemodynamic changes. However, the process of monitoring hemodynamics during ductal closure (MHDC, i.e. the 'arch watch') is variable across institutions and can be insensitive to critical deficiencies in oxygen delivery in the setting of decreased blood flow, even in subspecialized ICU environments. Current approaches to monitoring hemodynamic changes in neonates with possible AAO revolve around non-invasive measurements of oxygen saturation (i.e. pulse oximetry, near infrared spectroscopy (NIRS)) and tissue perfusion (i.e. femoral pulse strength, urine output, blood pressure). There are no publications which systematically and concurrently assess these trends during this hemodynamic transition, and as such, there are no agreed upon thresholds to alert clinicians that a developing AAO is causing impaired tissue perfusion/oxygenation. Exploration of traditional measures of tissue oxygenation may prove more sensitive and specific at identifying compromise in newborns with critical AAO. For example, certain pulse oximetry waveform characteristics (photoplethysmography, PPG) have shown differences in healthy newborns versus those with CoA. Resonance Raman spectroscopy (RRS) is another validated non-invasive method that assesses peripheral tissue oxygenation in neonates and has been shown to correlate well with invasive markers of tissue oxygenation. The investigators and others have utilized RRS in healthy neonates and in animals to detect tissue hypoperfusion. To test the hypothesis that a validated MHDC process that combines commonly used non-invasive monitoring tools, new components of these traditional tools, and RRS, will have improved sensitivity in detecting critical impairments to tissue oxygen delivery in newborns with suspected critical AAO, the investigators identified the following aims:

Aim I: To assess the reliability of currently deployed non-invasive markers of tissue oxygenation/perfusion (femoral pulse strength, pre- vs. post- ductal blood pressure and saturation gradient, cerebral/renal NIRS, and urine output) in identifying a critical AAO that will need intervention in the newborn period.

Aim II: To explore the sensitivity of PPG to identify critical AAO requiring intervention in the newborn period.

Aim III: To determine the feasibility of assessing oxygen utilization at the tissue level based on RRS during MHDC and examine its predictive capability in identifying those infants with AAO who will require arch intervention in the newborn period.

ELIGIBILITY:
Inclusion Criteria:

* Infants with echocardiography-based possible or definite aortic arch obstruction and <1 month postnatal age admitted to the CICU
* Clinical team assent to approach family, (3) parent/guardian informed consent. Inclusion criteria includes infants with concurrent other congenital heart disease, or simple Coarctation of the aorta or arch hypoplasia

Exclusion Criteria:

* Known carrier status for resistant organisms. Resistant organisms are defined as MRSA and VRE.

Ages: 0 Days to 60 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants with prenatal or postnatal echocardiographic findings concerning for or diagnostic of aortic arch obstruction admitted to the BCH CICU.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with arch or CoA repair | First 3 postnatal months
  Surgical or catheter-based repair of the aortic arch or coarctation of the aorta

SECONDARY OUTCOMES:
Number of participants with echocardiographic finding of aortic arch obstruction | First 3 postnatal months
  Echocardiographic finding of aortic arch obstruction defined as blunted doppler in the descending aorta or presence of pathognomonic characteristic of CoA such as clear posterior shelf
Number of participants with end organ damage as evidence by necrotizing enterocolitis, or acute kidney injury in the first three postnatal months | First 3 postnatal months
  Necrotizing enterocolitis will be defined as the presence of pneumatosis intestinalis as documented in an attending-read radiology report. Acute kidney injury will be defined per modified neonatal KDIGO guidelines of stage I or greater AKI (serum creatinine SCr rise of greater than 0.3 mg/dL within 48 hours or SCr rise greater than 1.5-1.9x baseline SCr within 7 days) or if no creatinine data are present for the patient, then using urine output criteria of less than or equal to 1 ml/kg/hr of urine output for 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: John Kheir, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No